CLINICAL TRIAL: NCT05115383
Title: The Effects of Exercise and Training Status on the Counter-regulatory Axis of the Renin-angiotensin-system.
Brief Title: Effects of Exercise on the Renin-angiotensin System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 117957
Record Dates: First submitted 2021-10-03; First posted 2021-11-10 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedentary Group (Active Comparator): Individuals who are physically active for less than 75 minutes of moderate to vigorous physical activity a week will be placed in the sedentary group.
  Interventions: Other: VO2 Max test
- Active Group (Active Comparator): Individuals who are physically active for greater than 150 minutes of moderate to vigorous physical activity will be placed in the active group.
  Interventions: Other: VO2 Max test

INTERVENTIONS:
Other: VO2 Max test — The participant will be equipped with a vo2 mask or mouthpiece. They will get on the bike and begin with a 5 minute warmup ranging from 30-100 watts. After the warm up there will be a 15-30 watt increase every minute in the cadence that the participant is required to maintain. Once the participant has decided to stop pedalling, the participants mask will be removed to ensure they are feeling well. They will allowed to continue pedaling at their own pace for a cool down for up to two minutes.

SUMMARY:
Angiotensin converting enzyme-2 (ACE2) is part of the renin-angiotensin system (RAS), which is involved in maintaining blood flow and electrolyte balance. It has been shown in obese and hypertensive individuals that levels of another molecule Angiotensin converting enzyme (ACE) are much higher, leading to inflammation, fibrosis, vasoconstriction and high blood pressure. ACE2 has a protective effect from ACE, leading to anti-inflammatory, anti-fibrotic and vasodilating effects.

In animal models, it has been shown that aerobic exercise can increase levels of ACE2, while decreasing levels of ACE and offers protection to the cardiovascular system by keeping these two molecules balanced. Although the effects of exercise on the classical arm of the RAS have been studied significantly, ACE2 is a relatively new discovery and has not been studied as extensively in humans. The purpose of this research is to determine the effects of exercise training status on the RAS, specifically on ACE2 and its products.

DETAILED DESCRIPTION:
The design of the proposed study is an intervention study, where participants are selected into either a physically active group or a sedentary group. The physically active group will be set as our control, as the physiological stress of the exercise protocol should be lower in the physically active group and limit the magnitude of the response. Both groups will be exposed to the same experimental procedure. Participants will be placed in their group based on their responses to the CSEP Get Active questionnaire. Individuals who do not accumulate less than 75 minutes of moderate to vigorous physical activity a week will be placed in the sedentary group, while those who accumulate more than 150 minutes will be placed in the active group.

Participants will be asked to avoid anti-Inflammatory medications, drugs, alcohol and smoking 48 hours prior to any of the sessions.

Participants in both groups will undergo the same testing procedure. Tests will include densitometry and a graded exercise test to measure maximum VO2 and associated parameters. Venipuncture (10 ml) will be performed before, after and 30 minutes post VO2 max test. The proposed study analysis will be conducted using a dependent groups ANOVA and Tukey's post hoc testing.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-39
* ability to exercise to exhaustion
* ability to give informed consent

Exclusion Criteria:

* chronic consumption of recreational drugs, tobacco or alcohol
* on any prescription medication or anti-inflammatory medications
* diagnosed with any chronic conditions
* current diagnosis with COVID-19
* BMI >30
* Engage in 75-150 minutes of moderate to vigorous physical activity a week

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-07-08 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in the mean response to an acute bout of physical activity in the components of the renin-angiotensin system | measurements will be taken before, immediately post and 30 minutes post exercise.
  Measurements of Angiotensin(1-10) and Angiotensin(1-9) will be analyzed using ELISA kits.

SECONDARY OUTCOMES:
Changes in the baseline measurements of the renin-angiotensin system between physically active and sedentary males. | Measurements will be made prior to commencement of exercise protocols.
  Ratios of Angiotensin(1-10) and Angiotensin(1-9) will be compared between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Nutrition Laboratory, Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided